CLINICAL TRIAL: NCT05543941
Title: Evaluating XPERIENCE™ Advanced Surgical Irrigation on Risk of Periprosthetic Joint Infection: A Multicenter Randomized Controlled Trial
Brief Title: Evaluating XPERIENCE™ Advanced Surgical Irrigation
Acronym: XPERIENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Next Science TM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISR-0104
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hip Osteoarthritis; Hip Arthritis; Knee Osteoarthritis; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- XPERIENCE Advanced Surgical Irrigation (Experimental): Patients will receive the XPERIENCE Advanced Surgical Irrigation prior to wound closure.
  Interventions: Device: XPERIENCE Advanced Surgical Irrigation
- Dilute Betadine (Active Comparator): Patients will receive Dilute Betadine solution prior to wound closure.
  Interventions: Device: Dilute Betadine

INTERVENTIONS:
Device: XPERIENCE Advanced Surgical Irrigation — The patient will undergo THA, TKA, or HR with irrigation of the deep wound prior to fascial closure consisting of XPERIENCE Advanced Surgical Irrigation (XP). XP solution will be applied prior to fascial closure and left to soak for up to 3 minutes. Remaining product will be suctioned away throughout the procedure. No rinsing should take place after irrigation and surgical site will be closed according to site standard operating procedures.
  Other Names: XP
  Arms: XPERIENCE Advanced Surgical Irrigation
Device: Dilute Betadine — The patient will undergo THA, HR or TKA with irrigation of the deep wound prior to fascial closure consisting of Dilute Betadine (DB). DB concentration will be standardized at 0.3% povidone-iodine. DB will be prepared by combining 30 mL of sterile 10% povidone-iodine (from a sterile catheter pack) with 1 L of 0.9% saline in a sterile splash basin. Solution will be left to soak for up to 3 minutes and remaining povidone-iodine solution will be suctioned away. Area will then be rinsed with 1L of normal saline. Surgical site will be closed according to site standard operating procedures.
  Other Names: DB; Providone-Iodine
  Arms: Dilute Betadine

SUMMARY:
A prospective, multi-center, double-arm, parallel, interventional, randomized, controlled clinical trial to assess the rate of periprosthetic joint infection (PJI) in patients undergoing primary total knee arthroplasty (TKA), total hip arthroplasty (THA) or hip resurfacing (HR) with XPERIENCE™ (XP) Advanced Surgical Irrigation versus dilute Betadine (DB).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or older
2. Diagnosis of osteoarthritis, inflammatory arthritis, osteonecrosis, or post-traumatic arthritis to the affected joint.
3. Primary TKA, THA, and HR
4. Subjects receiving both cemented or uncemented orthopaedic implants
5. Willing and able to sign written consent, follow study protocol and attend follow-up

Exclusion Criteria:

1. Inability or refusal to sign informed consent form
2. Non-English or French speaking, and no licensed translator, family member or substitute decision maker available.
3. Prior arthroplasty procedure to the affected joint
4. Procedures involving solid HA implants
5. Oncologic diagnosis to the affected joint.
6. Non-TKA, THA or HR prosthesis (i.e., hemiarthroplasty, unicompartmental arthroplasty etc.)
7. Allergy to any of the components of XP Advanced Surgical Irrigation
8. Allergy to iodine
9. Presence of concurrent active infection, primary immunodeficiency, history of uncontrolled HIV (CD4 count <200 cells/uL), treatment with immunomodulatory medications for malignancy or autoimmune disease (with exception to inflammatory arthritis), chronic glucocorticosteroid use (≥20 mg of prednisone daily for at least 1 month with another cause of immunosuppression), and solid organ and/or bone marrow transplantation.
10. History of septic arthritis to the affected joint within two years of surgery(1).
11. History of steroid injection to the affected joint within the three months preceding surgery.
12. Simultaneous bilateral total joint arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7600 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of acute (<90 days post-surgery) PJI | 2 weeks after surgery, 3 months after surgery, within 90 day of surgery
  Number of patients diagnosed with periprosthetic joint infection as per the diagnostic criteria outlined by the 2018 International Consensus Meeting of the Musculoskeletal Infection Society for Acute PJI.

SECONDARY OUTCOMES:
Rate of Superficial Wound Infections | 2 weeks after surgery
  Number of superficial wound infections
Rate of PJI at 1 year | 12 months after surgery
  Number of patients diagnosed with periprosthetic joint infections at 1 year after surgery
Subgroup analysis of PJI rates for high-risk patients | 3 months after surgery, 12 months after surgery
  Number of patients diagnosed with PJI at 3 months and 1 year in higher risk patient categories (morbid obesity (BMI >40kg/m2), diabetes mellitus, chronic kidney disease, inflammatory arthritis, active smokers (nicotine))
Patient Reported Functional Outcome Scores | Before surgery, 3 months after surgery, 12 months after surgery
  As measured by the Oxford Hip Score (OHS) or Oxford Knee Score (OKS)
Patient Reported Quality of Life Scores | Before surgery, 3 months after surgery, 12 months after surgery
  As measured by the Patient-Reported Outcomes Measurement Information System (PROMIS)
Wound Complications (non-infection) requiring revision surgery | 2 weeks after surgery
  Number of patients requiring a revision surgery for a non-infection related wound complication

CONTACTS AND LOCATIONS:
Overall Officials: Simon Garceau, MD, Principal Investigator — The Ottawa Hospital
Locations (9):
- Canada (9):
  - University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Center, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Humber River Health, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - CHU de Quebec-Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available to other researchers